CLINICAL TRIAL: NCT03626402
Title: End-of-Life Care for African Americans: An Outpatient Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ramona L. Rhodes, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU 042016-050; CCCDA-16-003-01 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2017-02-17; First posted 2018-08-13 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Advance Care Planning
Keywords: advanced cancer; African American

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing an intervention group to usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): These patients will be exposed to the educational intervention, including viewing the video, "Planning for the Care You Want," and meeting with a lay health advisor to discuss advance care planning and initiate plans, as patients wish.
  Interventions: Behavioral: Planning for the Care You Want
- Control - Usual Care (No Intervention): These patients will not be exposed to the educational intervention and will receive usual care. All patients will be mailed an informational brochure about advance care planning with a reminder letter two weeks after completing their baseline survey.

INTERVENTIONS:
Behavioral: Planning for the Care You Want — 25-minute culturally specific educational video informing viewers about advance care planning options, palliative care, and hospice care and meeting with a lay health advisor to discuss content of the video.
  Arms: Intervention

SUMMARY:
Racial differences in health care are documented across the health care continuum and persist in aging and end-of-life (EOL) care. African Americans (AA) and other underrepresented minorities often choose more aggressive therapies in the terminal stages of illness. Main reasons for these EOL disparities include: lack of knowledge of and misperceptions about palliative and hospice care, spiritual beliefs, and mistrust in the health care system. Despite the presence of national hospice guidelines, interventions addressing these disparities have been limited and often not rigorously evaluated. Most interventions to promote EOL care were done in majority populations and focused predominantly on trying to change physician awareness of patient's pain, symptoms, and values or to change physician communication behavior. While these early studies made tremendous contributions to the study of EOL care and the needs of the terminally ill, the interventions associated with these studies did not reach their desired effectiveness. The investigator proposes an innovative strategy that would focus specifically on previously identified physician and patient barriers to utilization of advance directives, palliative care, and hospice care among AA cancer patients. The goal of this patient-centered project is to increase the awareness of and willingness to discuss EOL care options among AAs with metastatic cancer. To overcome the dual challenges of physicians' difficulty with prognostication and reluctance to discuss EOL care, the investigator will harness data in the electronic medical record (EMR) to automatically identify AA patients with metastatic breast, lung, colorectal, prostate and other serious cancer who are eligible for counseling about palliative and EOL care options. To change AA patients' knowledge and attitudes toward palliative and EOL care options, and address issues of medical mistrust, the investigator will design and pilot test a culturally sensitive, patient-targeted intervention that will combine multimedia materials and a culturally concordant lay health advisor (LHA) who will deliver tailored education and counseling. The investigator has chosen a LHA delivery strategy because past studies have shown that they are best suited to address medical mistrust and perceived conflict between spiritual beliefs and health care decisions.

DETAILED DESCRIPTION:
The investigator proposes a three-phase project to improve awareness of use of advance directives, palliative care and hospice services among patients with metastatic cancer by creating and evaluating a multifaceted culturally sensitive intervention that targets specific previously identified barriers to EOL care for AAs, including: knowledge, attitudes, and awareness of options for care, conflict between patients' spiritual beliefs, and the general hospice and palliative medicine philosophy of care, and medical mistrust. Aim 1 will refine and validate the e-EOL computerized algorithm to identify persons with stage III and IV breast, lung, colorectal, or other serious cancer who are appropriate candidates for discussions about advance care planning, palliative care, and hospice in the outpatient setting. The work in Aim 1 seeks to overcome the upstream barrier that physicians often have difficulty with prognostication and are reluctant to discuss prognosis and EOL care options with patients. Aim 2 will involve continued stakeholder engagement and the conduct of focus groups with oncologists and primary care providers at Parkland Hospital and its affiliated clinics to determine how to make the intervention feasible and acceptable to patients, caregivers, and providers. The investigator also will obtain feedback on our newly developed video and written educational materials that communicate key messages about EOL care options and overcome common barriers. In Aim 3, the investigator will test the preliminary feasibility, acceptability, and efficacy of the intervention that uses the e-EOL algorithm to identify AA patients with advanced cancer who are eligible for care discussions and then deploy a culturally concordant behavior change intervention that combines a Lay Health Advisor (LHA) and video and written materials. Use of an LHA will help overcome the providers' reluctance or lack of time to discuss EOL care issues and mitigate medical mistrust. The three linked studies provide the necessary sequence of research projects and multidisciplinary learning experiences needed to accomplish the PI's scientific and training goals. It will also lay the groundwork for a fully powered RCT to test the efficacy of a multifaceted EOL care counseling intervention vs. usual care.

Details of Research Design and Methods for Aim 1: Refine an e-EOL algorithm to identify patients with metastatic cancer in the outpatient setting. Aim 1 will expand and validate the e-EOL algorithm to identify patients with advanced cancer who are appropriate candidates for discussions about EOL care options in the outpatient setting. The e-EOL algorithm will assist physicians with determining prognosis more accurately and will provide a mechanism for systematically identifying candidates for a subsequent EOL care counseling intervention outlined in Aim 3.

Details of Research Design and Methods for Aim 2: The investigator will refine components of a culturally sensitive intervention to improve knowledge of and intent to consider EOL care options. Use of decision aids, educational videos, and LHAs has been shown to be effective in improving medical knowledge and shared decision making and reducing racial disparities for several clinical conditions. Though there have been few applications of these promising approaches to palliative and EOL care, recent use of decision aids in improving knowledge about the goals of care for persons with advanced dementia, have shown promise. Aim 2 will iteratively refine the intervention messages delivered through a combination of novel DVD segments that we have developed, print materials, and guided discussions by a culturally concordant LHA. Through qualitative methods, the team will test the language, framing, and communication strategies for conveying intervention messages and obtain feedback from primary care and oncology providers at Parkland Hospital to verify the appropriateness of these messages as intended by investigators.

Details of Research Design and Methods for Aim 3: Assess the feasibility and acceptability of a multifaceted EOL care behavior change pilot intervention. The pilot intervention will combine the refined elements from Aims 1 and 2, to conduct a small pilot RCT comparing the intervention group to a usual care control group. All of these aims taken together lay the groundwork for a future, fully powered RCT.

Description of the Pilot Intervention: The EOL LHA will meet with eligible patients and their caregivers to tell them their doctor approved of them receiving more information about their treatment options. The LHA will then assist the eligible patients and caregivers in watching the EOL care DVD segments (the video modules described in Aim 2 targeted to their pre-intervention survey needs assessment). After the patients and caregivers watch the DVD, the LHA will answer questions and provide additional information. They will then use counseling scripts created by the PI and research team to probe in more depth the patient's goals of care, and understanding of their clinical condition, prognosis, and treatment options. They will tailor the discussion to the patient's values, preferences, concerns, and clinical circumstances. Those who express interest in hearing more about EOL care options will be encouraged to discuss this with their doctor. The counselor will offer to update their physician on their discussion and help communicate the patient's desire for a palliative care consult or advance directive (if that is something they wanted). Specific questions about prognosis will be referred to the treating physician. Formal palliative care referrals will be ordered and performed in the usual fashion with the exception that the patient may ask the LHA to update the palliative care team on their prior discussions, concerns, and preferences. The LHA will follow up with patients the day after they view the educational video to answer any additional questions and again within one week to assist patients with advance care planning questions and referrals. All intervention sessions will be audiotaped to ensure intervention fidelity.

Usual Care: Participants randomized to usual care will proceed with clinical care as already routinely implemented by their physicians. At the time of recruitment, they will be asked to identify their primary caregiver who will also be contacted. Patient-caregiver pairs who are randomized to usual care will also be asked if they would be willing to be contacted at 1, 3 and 6-month intervals to complete the post-study assessment. All participants will be mailed a reminder letter that study staff will be contacting them to participate in follow-up surveys a couple of weeks prior to the 1-month surveys. The reminder letter will include an informational brochure that briefly and simply summarizes advance care planning options.

Primary Outcomes: Feasibility and acceptability are the main process outcomes. Feasibility is success in accurately identifying eligible patients via the e-EOL algorithm (number flagged, specificity, positive predictive value), and numbers and rates of patients completing the pilot intervention and follow-up interviews. Acceptability will be measured with Likert scale items rating "understandability, informativeness, balance, right amount of information, helpfulness, and "recommending this to others" used in published trials of decision aids. The LHA will also ask open-ended questions on things patients did or did not like about the intervention. The primary decision making outcome is change in intent to discuss EOL care options based on the Transtheoretical Stages of Change Model, an approach used in many other realms. The investigator will categorize patients into the following stages: 1) Pre-contemplation: is unaware of EOL care options/has not thought about discussing this with a provider; 2) Contemplation: is aware of EOL care options/thinking about discussing options; 3) Preparation: intends to discuss EOL care issues with the doctor/has a plan for talking about it; 4) Action: has a discussion with the provider about EOL care. The completion stage is not applicable in this medical situation because the goal of the intervention is for the patient to have an informed discussion about benefits and harms of all treatment options including EOL care. The intent is NOT to get all patients to choose palliative care or hospice, or complete and an advance directive, but for them to understand how palliative care may benefit them now or in the future, and how it can be combined with curative care. The goal is for the patient to make "the right decision for them" based on knowing all of the facts and options.

Secondary Outcomes will measure: 1) Knowledge of prognosis and EOL care options: will be measured by a questionnaire from prior NCI-funded palliative care studies; 2) Decisional conflict will be assessed by the Decisional Conflict Scale, a validated 16 item scale measuring uncertainty about the best course of action and factors contributing to uncertainty. Scores <25 (on this 100-point scale) are associated with implementing decisions, and scores >38 with decisional delay; 3) Quality of life (QOL): will be assessed with the McGill QOL Questionnaire, a well-validated 20-item scale developed to measure QOL at the EOL; 4) Healthcare utilization will include: outpatient visits (incl. palliative care), ED visits, hospitalizations, total hospital days, and use of hospice services (type and time to hospice initiation); 5) Date and place (hospital, hospice, home) of deaths within a 6 month follow-up period will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. breast, lung, colon, prostate or other advanced cancer diagnosis
2. English proficient
3. African American
4. mentally competent

Exclusion Criteria:

1) not currently receiving palliative or hospice care

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of relying upon the intervention algorithm to identify eligible patients | This will be assessed from the time of initiating patient recruitment (April 2017) through completion of recruitment of new patients (April 2018), up to 56 weeks.
  This will be assessed by the principal investigator reviewing the medical records of patients flagged by the algorithm as eligible for participation to verify their eligibility and confirming those who meet study inclusion criteria.
Acceptability of intervention among patients randomized to the intervention arm | Assessed at the end of the intervention, which occurs approximately two weeks after the baseline survey with those patients randomized to receive the intervention. This will be assessed beginning in April 2017 and ending in April 2018, up to 52 weeks.
  Patient acceptability will be determined by the lay health advisor asking the patient, "Is this video something that you would recommend that your family and/or friends watch?" Responses will be noted "yes, no, refused, or don't know." Then they will be asked, "Why/why not?" and their responses written verbatim.
Participant change in intent to discuss EOL care options | Assessed at baseline and at 1, 3, and 6 months of baseline beginning April 2017 and ending October 2018, up to 78 weeks.
  Changes in intention to discuss EOL care options will be assessed for all patients in both arms of the study by using the Transtheoretical Stages of Change Model.

SECONDARY OUTCOMES:
Knowledge of prognosis and EOL care options | Assessed at baseline and at 1, 3, and 6 months of baseline beginning April 2017 and ending October 2018, up to 78 weeks.
  Knowledge of prognosis and EOL care options will be measured by using survey questions designed to assess this.
Decisional conflict about preferences for EOL care | Assessed at baseline and at 1, 3, and 6 months of baseline beginning April 2017 and ending October 2018, up to 78 weeks.
  Decisional conflict will be assessed by using the Decisional Conflict Scale, a validated tool for scoring uncertainty related to decision making. Patients are asked, "If the doctors told you that your illness could not be cured, which treatment option would you prefer?" Patients must choose one of three choices: 1) "All treatment options available to help me live for as long as possible"; 2) "Palliative care"; or 3) "Hospice." They are then asked 10 follow-up questions to assess their certainty about their choice. The response choices to these 10 questions are "yes," "unsure," or "no." Each response choice is assigned a numeric value, 0, 2, and 4, respectively. The patient's total score is calculated by adding the values for all 10 questions, dividing the sum by 10, then multiplying that figure by 25. The patient's uncertainty score is calculated by adding the values of their responses to questions 9 and 10, dividing by 2, and multiplying that value by 25.
Participant perceptions about their quality of life | Assessed at baseline and at 1, 3, and 6 months of baseline beginning April 2017 and ending October 2018, up to 78 weeks.
  Perceptions of quality of life will be assessed by using the McGill Quality of Life Questionnaire-Revised (MQOL-R), a validated scale to measure the patient's perception of quality of life over the last two days. This instrument includes 15 questions to which patients respond with a number ranging from 0 to 10. For each question, the patient is told what a 0 means and what a 10 means--the definitions vary from question to question. For some questions, a 0 means "very bad" while a 10 means "excellent." For other questions, a 0 means "not a problem" while a 10 means "a tremendous problem." Patients can also refuse to answer or reply that they do not know.
Patient healthcare utilization | Assessed at 1, 3, and 6 months of baseline beginning May 2017 and ending October 2018, up to 74 weeks.
  Patient healthcare utilization will be assessed by research staff conducting chart reviews following each survey interval to quantify emergency department visits and hospitalizations, referrals to palliative care or hospice, and whether or not a patient has completed an advance directive following study initiation.
Date and place of death | Assessed at 1, 3, and 6 months of baseline beginning May 2017 and ending October 2018, up to 74 weeks.
  While conducting scheduled chart reviews, research staff will document the date and place (hospital, hospice, or home) if the medical record indicates that the patient is deceased.

CONTACTS AND LOCATIONS:
Overall Officials: Ramona L Rhodes, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT03626402/Prot_SAP_002.pdf
  • Informed Consent Form (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT03626402/ICF_003.pdf